CLINICAL TRIAL: NCT02375659
Title: Black Patients' Lived Experiences and Perceptions of Skin of Color Clinics
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: University of Wisconsin, Stout (Other)
Responsible Party: Principal Investigator, Stavonnie Patterson, Assistant Professor in Dermatology, Northwestern University
Other Study IDs: SSLP100114
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Perception of Skin of Color Clinics in African Americans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Focus group: Each focus group (4 total) will be approximately 90 minutes in duration. A trained facilitator will pose 8 scripted questions to the focus group participants and manage the conversation, ensuring all participants have an opportunity to respond and steering the conversation to remain on task. A note-taker will also be present at the focus group to document via handwritten notes the flow and content of the focus group conversation. All focus groups will be audio taped and transcribed.

SUMMARY:
Across the U.S. Skin of Color (SOC) clinics have been established with the goal of providing medical care and supporting research related to patients with skin of color. There have been no formal studies evaluating why patients seek medical care at SOC clinics or treatment outcomes. Reasons may include past experiences with other providers, the perception that providers working in these clinics have a special interest or knowledge in caring for patients with skin of color and thus may provide better care, the expectation of cultural sensitivity, the hope that their provider may have a similar ethnic background, and/or ease of communication with their provider. Through focus group discussions we aim to identify the factors influencing a patient's choice to seek medical care at a SOC clinic and to gain insight into the presence and impact of racial concordance between provider and patient. The current study will focus on self-identified African American patients with interest in conducting similar sessions with patients of other ethnicities and races in the future.

ELIGIBILITY:
Inclusion Criteria:

* Evaluated in the Northwestern Center for Ethnic Skin between February 1, 2015 and February 1, 2016.
* Evaluated by Drs. Stavonnie Patterson or Roopal Kundu
* Age 18 or older
* Self identified as African American/Black
* All subjects must have given signed, informed consent prior to participation in study.

Exclusion Criteria:

* English speaking as interpreters not available
* Existing mental health conditions that may interfere with focus group discussion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African American patients evaluated at the Northwestern Center for Ethnic Skin
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Common thematic responses of discussion groups | 100 minutes
  Audiotapes of focus group discussions will be transcribed, and the transcripts will be analyzed via a 'long-hand' inductive approach by two dermatologists and one psychologist. For each of the 8 posed focus group questions, the reviewers will independently induce a common thematic response. Collectively, they will then compare their independently derived themes, identifying themes of agreement and disagreement. Areas of disagreement will be further reviewed until a mutually agreed upon final set of themes is identified. The raw data corresponding to the item in question will be classified according to its theme.

CONTACTS AND LOCATIONS:
Overall Officials: Stavonnie Patterson, MD, Principal Investigator — Northwestern University Feinberg School of Medicine; Kristina Gorbatenko-Roth, PhD, LP, Principal Investigator — University of Wisconsin, Stout; Neil Prose, MD, Principal Investigator — Duke University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Barr DA, Wanat SF. Listening to patients: cultural and linguistic barriers to health care access. Fam Med. 2005 Mar;37(3):199-204. PMID 15739136
- [Background] Beach MC, Gary TL, Price EG, Robinson K, Gozu A, Palacio A, Smarth C, Jenckes M, Feuerstein C, Bass EB, Powe NR, Cooper LA. Improving health care quality for racial/ethnic minorities: a systematic review of the best evidence regarding provider and organization interventions. BMC Public Health. 2006 Apr 24;6:104. doi: 10.1186/1471-2458-6-104. PMID 16635262
- [Background] Cooper LA, Roter DL, Johnson RL, Ford DE, Steinwachs DM, Powe NR. Patient-centered communication, ratings of care, and concordance of patient and physician race. Ann Intern Med. 2003 Dec 2;139(11):907-15. doi: 10.7326/0003-4819-139-11-200312020-00009. PMID 14644893
- [Background] Cooper-Patrick L, Gallo JJ, Gonzales JJ, Vu HT, Powe NR, Nelson C, Ford DE. Race, gender, and partnership in the patient-physician relationship. JAMA. 1999 Aug 11;282(6):583-9. doi: 10.1001/jama.282.6.583. PMID 10450723
- [Background] Majette GR. Access to health care: what a difference shades of color make. Ann Health Law. 2003;12(1):121-42, table of contents. PMID 12705206
- [Background] Michalopoulou G, Falzarano P, Arfken C, Rosenberg D. Physicians' cultural competency as perceived by African American patients. J Natl Med Assoc. 2009 Sep;101(9):893-9. doi: 10.1016/s0027-9684(15)31036-1. PMID 19806846
- [Background] Phillips KL, Chiriboga DA, Jang Y. Satisfaction with care: the role of patient-provider racial/ethnic concordance and interpersonal sensitivity. J Aging Health. 2012 Oct;24(7):1079-90. doi: 10.1177/0898264312453068. Epub 2012 Aug 6. PMID 22869897
- [Background] Sauaia A, Dellavalle RP. Health care inequities: an introduction for dermatology providers. Dermatol Clin. 2009 Apr;27(2):103-7, v. doi: 10.1016/j.det.2008.12.001. PMID 19254652